CLINICAL TRIAL: NCT02892825
Title: Impact of Music on Hypertension During Cataract Surgery Performed Under Topical Anaesthesia
Brief Title: Music Listening for Cataract Surgery
Acronym: MUSICATOP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: K150903; 2016-A00728-43 (Other: ANSM)
Record Dates: First submitted 2016-07-19; First posted 2016-09-08 (Estimated); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Cataract Surgery
Keywords: Music; cataract surgery; topical anaesthesia; anxiety; hypertension
MeSH Terms: conditions — Anxiety Disorders; Hypertension | interventions — Music Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- music group (Experimental): music listening
  Interventions: Other: Music
- no music group (Active Comparator): no music listening
  Interventions: Other: No Music

INTERVENTIONS:
Other: Music — headphones with music
  Arms: music group
Other: No Music — headphones without music
  Arms: no music group

SUMMARY:
The purpose of the study is to assess the effect of music therapy on anxiety and hypertension during cataract surgery procedures performed under topical anaesthesia.

DETAILED DESCRIPTION:
Cataract surgery is the most frequent surgical procedure performed in Europe, usually done under topical anaesthesia. Restlessness and hypertension are the most frequent medical complications during surgery, potentially leading to surgical complications. Since the surgery is ambulatory and requires the patient's cooperation, heavy intravenous sedation should be avoided. However, this procedure is stressful, with patients experiencing high anxiety due to being awake and aware of the procedure on their eye and equipment. Music therapy may be considered as a non-pharmacologic and non-invasive mean to reduce anxiety and therefore intra-operative hypertension. To assess the effect of music therapy on anxiety and hypertension during cataract surgery procedures under topical anaesthesia, investigators intend to perform a randomized controlled trial. Depending on the results of the study, music therapy may subsequently be replacing the usual premedication before surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective cataract surgery performed under topical anaesthesia

Exclusion Criteria:

* Non topical anaesthesia
* Non ambulatory surgery
* Communication difficulties including language barrier, and mental disorders
* Age<18yo
* Hearing impairment
* Uncontrolled hypertension

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 313 (Actual)
Dates: Start 2017-02-02 (Actual); Primary Completion 2018-07-25 (Actual); Study Completion 2018-07-27 (Actual)

PRIMARY OUTCOMES:
Hypertensive event | Intraoperative every 5 minutes
  Non invasive measure through blood pressure cuff

SECONDARY OUTCOMES:
Anxiety score before surgery | before surgery
  on a visual analogue scale
Anxiety score after surgery | after surgery
  on a visual analogue scale
Duration of surgery | after surgery
Intraoperative surgical complications | during surgery
  reported by surgeon

CONTACTS AND LOCATIONS:
Overall Officials: Manon Guisse, nurse, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Cochin Hospital, Paris, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Guerrier G, Bernabei F, Lehmann M, Pellegrini M, Giannaccare G, Rothschild PR. Efficacy of Preoperative Music Intervention on Pain and Anxiety in Patients Undergoing Cataract Surgery. Front Pharmacol. 2021 Sep 30;12:748296. doi: 10.3389/fphar.2021.748296. eCollection 2021. PMID 34658886
- [Derived] Guerrier G, Abdoul H, Jilet L, Rothschild PR, Baillard C. Efficacy of a Web App-Based Music Intervention During Cataract Surgery: A Randomized Clinical Trial. JAMA Ophthalmol. 2021 Sep 1;139(9):1007-1013. doi: 10.1001/jamaophthalmol.2021.2767. PMID 34323929